CLINICAL TRIAL: NCT07071116
Title: Seminar in Unwavering Empowering Presence Optimized for Rehabilitation Teams
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SUPPORT
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Communication
Keywords: Communication Skills Training (CST); Rehabilitation Professionals
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Licensed rehabilitation professionals (Other): Licensed rehabilitation professionals (e.g., physical therapists, occupational therapists, speech-language pathologists) employed at St. Jude Children's Research Hospital actively involved in the care of pediatric oncology patients who will participate in the CST intervention
  Interventions: Other: Communication skills training
- St. Jude Bereaved Parent Educators (Other): St. Jude Bereaved Parent Educators who have participated as an educator in at least one other institutional educational event and will facilitate the CST intervention
  Interventions: Other: Communication skills training-Facilitator

INTERVENTIONS:
Other: Communication skills training — See Detailed Description
  Other Names: CST
  Arms: Licensed rehabilitation professionals
Other: Communication skills training-Facilitator — See Detailed Description
  Other Names: CST-Facilitator
  Arms: St. Jude Bereaved Parent Educators

SUMMARY:
The goal of this study to test the feasibility, acceptability, and potential impact of a serious illness communication skills training (CST) tailored to rehabilitation professionals to improve their comfort and confidence in navigating difficult conversations with patients and families.

Primary Objectives:

Aim 1: To assess feasibility and acceptability of a multidisciplinary co-designed interactive CST program for rehabilitation professionals who care for children with serious illness and their families.

Aim 2: To characterize the potential impact of this CST intervention on pediatric rehabilitation professionals.

Secondary Objective:

Aim 3: To examine the perspectives of bereaved parent educators on participation in the implementation of communication training for rehabilitation professionals.

DETAILED DESCRIPTION:
The Communication Skills training (CST) will last approximately 3 hours. It will consist of three main components: Part 1 will begin with an introductory case of an emotional parent, then a brief didactic with a framework on responding to emotion, and end with rehab professionals actively practicing 'drills' using the framework for responding to emotion. Part 2 will be a panel of bereaved parents. Learners will be asked to think of questions to ask the parents in advance and will also be invited to ask questions that come to mind in the moment. Part 3 will be focused on sharing serious news, beginning with an introductory case of sharing cancer progression, followed by didactic teaching in a VitalTalk framework, 'REMAP,' for sharing serious news and eliciting goals/values. Leaders will then introduce role-play via a demonstration case. Next, learners will be divided into small groups for discussion and role-play, with a strong emphasis on principles of psychological safety and learner autonomy. and incorporates didactic instruction, experiential learning, and involvement of bereaved parent educators.

Demographic information will be collected for participating bereaved parent educators and rehabilitation professionals. Rehabilitation professionals will complete pre-intervention self-assessment surveys immediately prior to the educational intervention. Post-intervention self-assessment surveys will be administered immediately after completion of the intervention and 3-months post-intervention to assess for retention. Rehabilitation professionals and bereaved parent educators will also be interviewed about their experience following the intervention. The interviews will be done on an individual basis either virtually or in-person.

ELIGIBILITY:
Inclusion Criteria: Intervention Participants

* Licensed rehabilitation professionals (e.g., physical therapists, occupational therapists, speech-language pathologists) employed at St. Jude Children's Research Hospital actively involved in the care of pediatric oncology patients.
* Willingness to participate in the communication skills training (CST) intervention and associated study activities.

Inclusion Criteria: Intervention Facilitators

* St. Jude Bereaved Parent Educators who have participated as an educator in at least one other institutional educational event
* Willingness to facilitate the communication skills training (CST) intervention and complete associated study activities.

Exclusion Criteria: Intervention Participants

* Non-rehabilitation professionals
* Individuals unable to attend the CST intervention session.

Exclusion Criteria: Intervention Facilitators

* Individuals unable to attend the CST intervention session.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve a mean score ≥3 on the Feasibility of Intervention Measure (FIM) scale | Approximately 3 months post intervention
  Investigators will compute the mean Feasibility of Intervention Measure (FIM) score for each participant using the Feasibility of Intervention Measure (FIM) and report the proportion of participants who achieve a mean score ≥3. The Feasibility of Intervention Measure (FIM) is used to assess how feasible it is to implement a specific intervention. The FIM measure includes four itemized responses that are scored from one to five (1=Completely disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Completely agree) such that one represents the lowest possible mean score and five the highest possible mean score. It is scored by averaging the responses to each of the four questions. Higher scores indicate greater perceived feasibility of the intervention.
Proportion of participants who achieve a mean score ≥3 on Acceptability of Intervention Measure (AIM) scale | Approximately 3 months post intervention
  Investigators will compute the mean Acceptability of Intervention Measure (AIM) score for each participant and report the proportion of participants who achieve a mean score ≥3. The Acceptability of Intervention Measure (AIM) is a four-item scale used to assess the acceptability of an intervention. It is scored by calculating the mean of the responses to its four items, each measured on a 5-point Likert scale(1=Completely disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Completely agree). This results in a final score ranging from 1 to 5, with higher scores indicating greater acceptability.
Proportion of participants who achieve a mean score ≥3 on the Intervention Appropriateness Measure (IAM) scale | Approximately 3 months post intervention
  Investigators will compute the mean Intervention Appropriateness Measure (IAM) score for each participant and report the proportion of participants who achieve a mean score ≥3. The Intervention Appropriateness Measure (IAM) is a four-item scale used to assess the appropriateness of interventions by capturing individual perspectives on the alignment of the intervention with professional values and perceived efficacy in meeting patient needs. Each item is rated on a 5-point Likert scale (1=Completely disagree, 2=Disagree, 3=Neither agree nor disagree, 4=Agree, 5=Completely agree). The score is calculated by averaging the responses to all items. A higher score on the IAM indicates a stronger perception that the intervention is appropriate for the given situation and context.
Potential impact of this CST intervention on pediatric rehabilitation professionals | Prior to the start of the intervention (day 1) and at the end of study, approximately 3 months
  Investigators will calculate the proportions of participants who select "Agree" or "Completely agree" in both the pre- and post-intervention surveys and conduct statistical tests, such as Fisher's exact test or the Chi-square test, to determine whether the change in these proportions over time is statistically significant.

SECONDARY OUTCOMES:
Perspectives of bereaved parent educators on participation in the implementation of communication training for rehabilitation professionals. | Within 3 months post intervention
  Interviews will be conducted with bereaved parent educators following the intervention. Interviews will be recorded, transcribed, de-identified, and analyzed using content analysis, an inductive approach which may include memo-writing, codebook development, coding, reconciliation, and synthesis to identify patterns and themes that emerge from the interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Cowfer, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols